CLINICAL TRIAL: NCT04222998
Title: Impact of Home-based Growth Charts on Child Linear Growth in Indonesia
Brief Title: Home-based Growth Charts in Indonesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: The Abdul Latif Jameel Poverty Action Lab Southeast Asia (Unknown); Department of Foregin Affairs and Trade, Australia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-39613; 73494 (Other Grant/Funding Number: Department of Foreign Affairs and Trade, Australia)
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Child Growth
Keywords: Home-based growth charts; Child nutrition; Growth faltering; Stunting; Indonesia
MeSH Terms: conditions — Growth Disorders | interventions — House Calls; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Sub-villages ("dusun") will be randomly assigned to control and treatment group with around 740 caregiver-child (9-14 months) dyads in each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Household receives the home-based growth chart
  Interventions: Other: Home-based growth charts; Other: Home visits for baseline surveys; Other: Home visits for end line surveys; Other: Measurement of child's height-for-age and weight-for-age
- Control group (Active Comparator): Household does not receive the home-based growth chart
  Interventions: Other: Home visits for baseline surveys; Other: Home visits for end line surveys; Other: Measurement of child's height-for-age and weight-for-age

INTERVENTIONS:
Other: Home-based growth charts — The growth chart contains simple information of nutritious food, health, and sanitation information at the top and height chart is located at the bottom where caregivers can measure their child's linear growth. Growth charts will be installed in intervention group homes just after the baseline survey.
  Arms: Intervention group
Other: Home visits for baseline surveys — Households will be visited for baseline surveys.
Other: Home visits for end line surveys — Households will be revisited after 1 year of grace-period for baseline end line surveys.
Other: Measurement of child's height-for-age and weight-for-age — The child's height-for-age and weight-for-age will be measured for participating dyads at the time of the baseline and end line surveys.

SUMMARY:
The investigators developed a home-based growth chart that offers a simple and inexpensive way for caregivers to have access to simple health and nutrition information guided by behavioural economics analysis as well as to track their child's linear growth, empowering them to act to improve their child's nutrition. Results from a pilot study conducted in rural Zambia suggest that growth charts installed in homes can increase awareness and reduce early-life growth deficits, particularly among children experiencing growth faltering. The main objective of this study is to assess the impact and cost-effectiveness of growth charts through a cluster-randomized trial in Indonesia. The primary outcome is child height-for-age z-score.

DETAILED DESCRIPTION:
The study is divided into two phases. In the first phase, growth chart development activities will be conducted in two villages in each of Manggarai Timur and Trenggalek districts to ensure the chart design is compatible with the local context and chart information is understandable to caregivers. Focus group discussions (FGDs), key informant interviews (KIIs), and door-to-door user testing will be conducted in each village. Results from the FGDs and KIIs will inform a draft growth chart design that will then be user tested in 10 households in each village. Qualitative interviews will be conducted with each household approximately two weeks after chart installation to gather insights on the usability of the growth chart. The chart design will then be finalized for use in the second phase of the study.

In the second phase, 1,480 caregiver-child dyads will be recruited and enrolled in the study as part of a baseline survey. Dyads will be sampled using a two-stage procedure. 110 villages will be selected proportionate to national census population size. All sub-villages ("dusun") within selected villages will be randomly assigned into two groups: 1) Growth chart; and 2) Control. Eligible caregiver-child dyads with children between 9 and 14 months will be selected from each sub-village.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers must be 19 - 55 years old
* One child of either gender, 9-14 months old
* Caregiver can have other children
* Caregiver of any occupation and income level
* Live in Manggarai Timur and Trenggalek during inception

Exclusion Criteria:

-Caregivers with a cognitive disability

Ages: 9 Months to 14 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1487 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Child height for age z-score (HAZ) | 12 months
  Height/length data will be converted to height for age z-score (HAZ) using WHO (World Health Organization) growth standards.
Child stunting | 12 months
  Child stunting is defined as height for age z-score (HAZ) < -2

SECONDARY OUTCOMES:
Child weight for age z-score (WAZ) | 12 months
  Weight data will be converted to weight for age z-score (WAZ) using WHO growth standards.
Early child development (ECD) | 12 months
  ECD will be evaluated with the Caregiver Reported Early Childhood Development Instruments (CREDI) Long Form which assesses child cognitive, motor, language, and social-emotional development. It provides a global, population-level measure of ECD for children in the 0-3 age range. The long form has about 60 items coded as Yes=1, No=0 and Don't know=8. The CREDI Long Form creates domain-specific developmental scores.

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Rockers, ScD, MPH, Principal Investigator — BU School of Public Health
Locations (1):
- The Abdul Latif Jameel Poverty Action Lab Southeast Asia, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No